CLINICAL TRIAL: NCT05073107
Title: The Effect of An Artificial Intelligence ("AI") Mobile Dental Application ("Dental Monitoring") in the Promotion of Self-Administered Plaque Control: A Randomized Controlled Trial
Brief Title: The Effect of A Dental Application to Promote Self-Administered Plaque Control: A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/00520
Record Dates: First submitted 2021-09-02; First posted 2021-10-11 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-04

CONDITIONS: Periodontitis; Gingivitis; Plaque, Dental
Keywords: oral hygiene; periodontitis; dental informatics; dental technology; patient reported outcome measures
MeSH Terms: conditions — Periodontitis; Gingivitis; Dental Plaque

STUDY DESIGN:
Intervention Model Description: To investigate the feasibility of the usage of a mobile dental application in the self-administration of plaque control in a two (2) parallel arm study with 52 subjects (n = 52). The study will take place over 2 visits (within 35 days): Visit 1 and 2.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test: With Dental Monitoring (Experimental): Dental Monitoring ("DM") Kit + 2-month DM subscription
  Required to take intra-oral videos (which will be translated into photographs) using the DM application weekly and it will be monitored by the delegated team members:
  * Day 0 (To be taken at the clinic)
  * Day 7 (To be taken in the evening after brushing teeth)
  * Day 14 (To be taken in the evening after brushing teeth)
  * Day 21(To be taken in the evening after brushing teeth)
  * Day 28 (To be taken before study Visit 2)
  There is a window period of +1 day for the intra-oral videos.
  Interventions: Other: Mobile Dental Application, Dental Monitoring ("DM")
- Control: Without Dental Monitoring (No Intervention): No DM Kit

INTERVENTIONS:
Other: Mobile Dental Application, Dental Monitoring ("DM") — o The Test group will be required to take intra-oral videos (which will be translated into photographs) using the DM application weekly and it will be monitored by the delegated team members:
  * Day 0 (To be taken at the clinic)
  * Day 7 (To be taken in the evening after brushing teeth)
  * Day 14 (To be taken in the evening after brushing teeth)
  * Day 21(To be taken in the evening after brushing teeth)
  * Day 28 (To be taken before study Visit 2) There is a window period of +1 day for the intra-oral videos.
  Arms: Test: With Dental Monitoring

SUMMARY:
Randomized Controlled Trial: to investigate the feasibility of the usage of a mobile dental application in the self-administration of plaque control in a two (2) parallel arm study with 52 subjects (n = 52). The study will take place over 2 visits (within 35 days): Visit 1 and 2.

Prospective Open Cohort Study: Patients referred to the Periodontology Department will be invited to participate in the study during the Oral Hygiene Phase. Routine clinical indices will be recorded at Visit 1 and Visit 2 before active non-surgical periodontal treatment commences.

DETAILED DESCRIPTION:
Visit 1 (Week 0, Day 0): Start of Study

* Subjects: The periodontal patients who have a dental appointment scheduled in the National University Centre for Oral Health, Singapore and fulfil inclusion/exclusion criteria will be recruited into the study by the delegated study team members. After written informed consent has been obtained and all the standard dental practices such as collecting the Routine Clinical Periodontal Parameters for evaluation and providing Oral Hygiene Instruction are done by the blinded study team member(s) termed as the Examiner. After which, the Participants will be randomized into 2 groups by delegated study team members.
* There will be two groups:

  * Test (n = 26): Dental Monitoring ("DM") Kit + 2-month DM subscription
  * Control (n = 26): No DM Kit
* The Examiner will be either the Co-investigator or an oral hygiene therapist engaged to be on the delegated study team. The same single blinded Examiner will examine all the participants of the study at both Visits 1 and 2.
* Based on the design of the study, there will be no deviation from the standard periodontal treatment protocol and intervals between treatment for this group of patients in the public healthcare setting with the exception for the test groups whereby the usage of an additional DM application which will be evaluated in this study.
* The Test group will receive DM as an additional monitoring aid. The delegated study team members will guide the Test group to download the DM application onto their mobile device, provide them with a DM Kit including full instructions (verbal and instruction pamphlet).
* In addition, the Test group will be taught by the delegated study team members:

  1. How to pair up a DM Scanbox with your smartphone https://youtu.be/y-q9Z8JMbzo
  2. How to perform DM Scans with ScanBox https://youtu.be/YT859VMGL18
* The Test group will be required to take intra-oral videos (which will be translated into photographs) using the DM application weekly and it will be monitored by the delegated team members:

  * Day 0 (To be taken at the clinic)
  * Day 7 (To be taken in the evening after brushing teeth)
  * Day 14 (To be taken in the evening after brushing teeth)
  * Day 21(To be taken in the evening after brushing teeth)
  * Day 28 (To be taken before study Visit 2) *There is a window period of +1 day for the intra-oral videos.
* The Control group will monitor their own oral hygiene without any additional aids.
* All patients will be given a soft-bristled toothbrush, fluoridated toothpaste and inter-dental aids by the delegated study team members. They will be instructed not to use any forms of mouth rinse.

Visit 2 (Week 4, Day 28 to Day 35): End of Study

* This visit will be between Day 28 and 35.
* The Test group will be given a short questionnaire by delegated study team members to evaluate their perspective on the "ease of use" and "satisfaction" using DM.
* The same Routine Clinical Periodontal Parameters clinical parameters will be measured again by the same blinded Examiner in Visit 1 and the clinical parameters evaluated.
* At the end of Visit 2, the subject will need to return the DM Kit during this visit. There is no more post follow up for this study and patient will continue with their next scheduled dental appointment by their primary care team.
* The delegated study team will collect the data from the Routine Clinical Periodontal Parameters (Full Mouth Periodontal Probing Depth, Bleeding on Probing, Recession and Plaque Index) that have been recorded at Visit 1 and Visit 2 for the following:

  * Primary Outcome: Difference in Full Mouth Plaque Score (%)
  * Secondary Outcomes: Participants' experience/feedback in the Test group on the use of the Dental Monitoring application.
* The delegated study team will analyze the photographs taken by the DM application and the data collected via the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 21 and 65 years old
2. Dentate patients
3. English speaking and literacy for verbal instructions including the usage of the DM application
4. Have access or own a smartphone with wifi and/or cellular connectivity
5. Ability to provide informed consent to participate in the study and willing to download the DM application onto their smartphone
6. Able to link and register their email account to receive notifications from DM application during the study

Exclusion Criteria:

1. Patients below 21 years old
2. Patients who is in dental pain
3. Patients with dementia
4. Patients who has compromised manual dexterity
5. Patients who had received Scaling and Polishing less than one month prior to examination and treatment
6. Pregnant or lactating women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Full Mouth Plaque Score (%) | Between Visit 1 (Day 0) and Visit 2 (between Day 28 and 35)
  Difference in Full Mouth Plaque Score using the disclosing two tone liquid by Curaprox
Full Mouth Bleeding Score (%) | Between Visit 1 (Day 0) and Visit 2 (between Day 28 and 35)
  Difference in Full Mouth Bleeding Score using a UNC periodontal probe, 6 surfaces per tooth (mesio-buccal, mid buccal, disco-buccal, mesio-lingual, mid-lingual and ditto-lingual) will be measured

SECONDARY OUTCOMES:
Satisfaction and Ease of Usage of the Dental Monitoring Application/Kit | At the end of Visit 2 (between Day 28 and 35)
  Participants' experience/feedback in the Test group on the use of the Dental Monitoring application.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Hui Fu, Dr, Principal Investigator — National University Centre for Oral Health
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Impellizzeri A, Horodinsky M, Barbato E, Polimeni A, Salah P, Galluccio G. Dental Monitoring Application: it is a valid innovation in the Orthodontics Practice? Clin Ter. 2020 May-Jun;171(3):e260-e267. doi: 10.7417/CT.2020.2224. PMID 32323716
- [Background] Chen YW, Stanley K, Att W. Artificial intelligence in dentistry: current applications and future perspectives. Quintessence Int. 2020;51(3):248-257. doi: 10.3290/j.qi.a43952. PMID 32020135
- [Background] Talla PK, Levin L, Glogauer M, Cable C, Allison PJ. Delivering dental care as we emerge from the initial phase of the COVID-19 pandemic: teledentistry and face-to-face consultations in a new clinical world. Quintessence Int. 2020;51(8):672-677. doi: 10.3290/j.qi.a44920. PMID 32778857
- [Background] Schwendicke F, Samek W, Krois J. Artificial Intelligence in Dentistry: Chances and Challenges. J Dent Res. 2020 Jul;99(7):769-774. doi: 10.1177/0022034520915714. Epub 2020 Apr 21. PMID 32315260
- [Background] da Costa CB, Peralta FDS, Ferreira de Mello ALS. How Has Teledentistry Been Applied in Public Dental Health Services? An Integrative Review. Telemed J E Health. 2020 Jul;26(7):945-954. doi: 10.1089/tmj.2019.0122. Epub 2019 Oct 1. PMID 31573410
- [Background] Avula H. Tele-periodontics - Oral health care at a grass root level. J Indian Soc Periodontol. 2015 Sep-Oct;19(5):589-92. doi: 10.4103/0972-124X.157875. PMID 26644730